CLINICAL TRIAL: NCT02969057
Title: Effects of Liquid Oil vs Oleogel Co-ingested With a Carbohydrate-rich Meal on Human Blood Triglycerides, Glucose, Insulin and Appetite.
Brief Title: Palm And Rice Bran Oil Study
Acronym: PARBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: University of Guelph (Other)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principle Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016/00932
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Glucose Response
Keywords: Lipidemic Response
MeSH Terms: interventions — Breakfast; Rice Bran Oil; Palm Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Breakfast only (No Intervention): Control breakfast providing 50g carbohydrate
- Breakfast with rice bran oil gel (Active Comparator): Control breakfast, plus 25g rice bran oil gel (solid)
  Interventions: Other: Breakfast with rice bran oil gel
- Breakfast with rice bran oil (Active Comparator): Control breakfast, plus 25g rice bran oil (liquid)
  Interventions: Other: Breakfast with rice bran oil
- Breakfast with palm oil gel (Active Comparator): Control breakfast, plus 25g palm oil gel (solid)
  Interventions: Other: Breakfast with palm oil gel
- Breakfast with palm oil (Active Comparator): Control breakfast, plus 25g palm oil (liquid)
  Interventions: Other: Breakfast with palm oil

INTERVENTIONS:
Other: Breakfast with rice bran oil gel — 25 grams of rice bran oil gel
  Arms: Breakfast with rice bran oil gel
Other: Breakfast with rice bran oil — 25 grams of rice bran oil
  Arms: Breakfast with rice bran oil
Other: Breakfast with palm oil gel — 25 grams of palm oil gel
  Arms: Breakfast with palm oil gel
Other: Breakfast with palm oil — 25 grams of palm oil
  Arms: Breakfast with palm oil

SUMMARY:
The objective of the present study is to compare the effects of liquid or solid state of food on glycaemia, lipaemia and insulinaemia. 25 participants aged between 21 and 45 years will be recruited from the general public in Singapore. Fingerpricks and cannulation may cause minor discomfort and there may be some slight bruising around the site. Fingerpricks and cannulation will be done by an experienced research nurse or a trained research officer to minimize participant discomfort. If bruising does occur, it should disappear within one day and it should not affect participants' regular daily activity. Participants will be limited to a maximum of one test per week. In addition, blood collection will be carried out in a sterile designated area and thus the risk of infection will be very low. On rare occasions, participants may feel unwell during or after the testing session. We have several metabolic suites with beds for these individuals to rest on. The research nurse and research officers will monitor the individuals' condition and they will be provided with a ride home if required. All the study foods will be prepared in a hygienic manner in a purpose-built research kitchen maintained to the highest hygiene standards. The research staff has undergone basic training in food hygiene procedures. Hence, the risk of infective acute gastroenteritis will be minimal. Participants will be provided with some snacks at the end of each testing session. They will also be reimbursed to compensate for their time and costs associated with travel and parking at the completion of the study. In addition, participants will be provided with their blood glucose, blood pressure, and body composition results, with a brief interpretation of these at the conclusion of the study.

DETAILED DESCRIPTION:
Design: This will be a randomised, crossover study with five sessions in total. 1.) Instant rice porridge with orange juice, 2.) Instant rice porridge with palm oil, with orange juice 3.) Instant rice porridge with palm oleogel, with orange juice 4.) Instant rice porridge with liquid rice bran oil, with orange juice 5.) Instant rice porridge with rice bran oleogel, with orange juice

Study population: Healthy Chinese males (BMI 18-25 kgm-2) with body weight >/=45 kg, aged 21-45 years with normal fasting blood glucose (<6.0 mM), will be recruited from the general public in Singapore. The exclusion criteria are people with major chronic disease such as heart disease, cancer or diabetes mellitus, glucose-6-phosphate dehydrogenase (G-6-PD) deficiency, glucose intolerance, intolerances or allergies to test products, as well as individuals who are taking insulin or drugs known to affect glucose metabolism. People with a major medical or surgical event requiring hospitalization within the preceding 3 months, individuals with the presence of disease or drugs which influence digestion and absorption of nutrients, people who are on any therapeutic diet/ drug therapy and smokers will be excluded.

Screening visit: During the screening session, participants will receive an informed consent form and given ample time to go through it and rectify any queries they have. If they decide to take part in the study, they will be asked to sign the informed consent form. They will then be asked to complete a screening questionnaire, baseline measurements including anthropometric measurements, blood pressure, and physical activity level will be collected from each participant in order to determine their eligibility. Body weight and body composition will be measured using bioelectrical impedance analysis. Height will be measured using a stadiometer in order to calculate participants' BMI. Blood pressure will also be measured. All measurements will be taken in duplicate. Participants will then be scheduled for the 5 subsequent test visits. The screening visit will take approximately 1 hour.

Screening questionnaire: The screening questionnaire will include contact information, demographic, general health details, and physical activity level. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes. Physical activity level will be measured using a previously validated international physical activity questionnaire.

Meal composition: The test meal will consist of cooking oil (palm oil or rice bran oil in either liquid or gelled form made with ethylcellulose), orange juice and commercially available instant porridge.

Test visits: During the testing sessions, participants' glycaemic, insulinaemic, and lipaemic responses to the test meals will be measured. Participants' metabolic satiety for the test meals will also be assessed at regular intervals throughout the testing session. The test duration for each treatment is 6.5 hours and the testing sessions will take place at least 1 week apart. Subjects will be instructed to avoid strenuous physical activity for at least 3 days and avoid caffeine and alcohol consumption for at least 1 day prior to visiting the CNRC for their study trials. Participants will be asked to standardise their diets and to refrain from alcohol and exercise the day before their testing sessions. At the beginning of the testing session, a cannula will be inserted into participants' arms. One fasting blood sample will be collected by fingerprick and venous cannulation. A drop of blood will be collected into a HemoCue® cuvette (Helsingborg, Sweden) for blood glucose analysis. In addition, 5 milliliters of venous blood will be collected into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA for the analyses of plasma triglyceride, insulin and non-esterified fatty acids concentrations. Participants will then consume treatment meal within 10 minutes. Blood samples will be taken at baseline, 10, 20, 30, 45, 60, 90, 120, 150 and 180, 210, 240, 270, 300, 330 and 360 minutes. The amount of blood that will be collected at every time point will be approximately 5 mL. A maximum of 16 blood samples for will be collected by fingerprick and cannulation. A total of 400mL approximately of blood will be taken for the study. Glycaemic, insulinaemic, and lipaemic responses will be determined using the method described by Wolever and Jenkins. The area under the curve will be determined as the area of those increments above baseline only.

Participants will also be asked to rate their 'liking' for the test meal. Participants will rate their 'overall liking' for the test meal on a 100 mm VAS anchored with 'dislike extremely' (0 mm), 'neither like or dislike' (50 mm) and 'like extremely' (100 mm) immediately after they consume the test meal. Metabolic satiety: On the testing session days, participants will be asked to record their appetite ratings on a 100 mm visual analogue scale (VAS) immediately before they consume the test meal, then at every 30 minutes interval as peak changes are usually observed at 15-30 minutes after a test meal, based on previous studies.. The appetite-rating questionnaire will include questions on hunger, desire to eat, prospective consumption, fullness, and preoccupation with thoughts of food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male
* Age between 21 and 45 years
* BMI 18-25 kg/m2
* Body weight >/=45 kg
* Normal Blood Pressure (=140/90 mmHg)
* Normal Fasting Blood Glucose (<6.0 mM)

Exclusion Criteria:

* People who take part in sports at competitive/endurance levels•
* People with major chronic disease such as heart disease, cancer or diabetes mellitus
* People who are glucose-6-phosphate dehydrogenase (G-6-PD) deficiency
* People who have intolerances or allergies to test products
* Individuals who are taking insulin or drugs known to affect glucose metabolism and body fat distribution
* People with a major medical or surgical event requiring hospitalization within the preceding three months
* Individuals with the presence of disease or drugs which influence digestion and absorption of nutrients
* People who are on any therapeutic diet/ drug therapy
* Smokers

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose over 180 minutes period | 180 minutes
  Blood obtained through fingerprick, analysed using Hemocue analyser.
Change in postprandial serum triglyceride over 360 minutes period | 360 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser. Venous plasma triglyceride will be assessed at 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180, 210, 240, 270, 300, 330 and 360 minutes
Change in postprandial serum glucose over 360 minutes period | 360 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser. Venous plasma triglyceride will be assessed at 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180, 210, 240, 270, 300, 330 and 360 minutes

SECONDARY OUTCOMES:
Change in postprandial plasma insulin over 360 minutes period | 360 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser. Venous plasma insulin will be assessed at 0, 10, 20, 30, 45, 60, 90, 120, 150 and 180, 210, 240, 270, 300, 330 and 360 minutes
Change in postprandial appetite over 360 minutes period | 360 minutes
  Appetite ratings will be assessed at 10, 20, 30, 45, 60, 90, 120, 150 and 180, 210, 240, 270, 300, 330 and 360 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- JeyaKumar Henry, Singapore, Singapore

REFERENCES:
- [Derived] Tan SY, Peh E, Siow PC, Marangoni AG, Henry CJ. Effects of the physical-form and the degree-of-saturation of oil on postprandial plasma triglycerides, glycemia and appetite of healthy Chinese adults. Food Funct. 2017 Dec 13;8(12):4433-4440. doi: 10.1039/c7fo01194f. PMID 29090299